CLINICAL TRIAL: NCT03923296
Title: PERTH 2: Co-design of a Home-based Monitoring Service for Cancer Patients, Carers and Health Care Professionals to Optimize Delivery of Systemic Therapy.
Brief Title: PERTH 2: Co-design of a Home-based Monitoring Service for Cancer Patients to Optimize Delivery of Systemic Therapy.
Status: Completed | Type: Observational
Sponsor: Entia Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: IRAS: 234137
Record Dates: First submitted 2019-04-16; First posted 2019-04-22 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Cancer
Keywords: point of care; home monitoring; device; blood
MeSH Terms: conditions — Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HCPs: Health care professional interviews (market research)
  Interventions: Behavioral: Interviews
- Patients or caregivers: Patients or caregivers interviews
  Interventions: Device: Blood measurement and monitoring; Behavioral: Interviews

INTERVENTIONS:
Device: Blood measurement and monitoring — Blood from a single fingerprick will be used to used to measure and monitor patients blood parameters.
  Groups: Patients or caregivers
Behavioral: Interviews — Focus group interviews

SUMMARY:
Iterative co-design study where patients receiving systemic cancer therapy, carers and healthcare professionals involved in delivering cancer therapy, work with Entia to design a home based blood monitoring service. The iterative process means that at each stage of the development process, Entia will be building on what is learnt in the previous stage.

DETAILED DESCRIPTION:
The study will use feedback provided by patients, carers and heatlhcare professionals to inform the changes that are necessary to develop a successful, user friendly home-based blood monitoring service for cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Adequate english to participate in focus groups and workshops without an interpreter
* Patients of the study site who are currently undergoing systemic therapy or have previously undergone systemic therapy within the past 12 months
* Patients willing to participate in at least 60-minute and ideally 90-minute workshops at the designated study location, time and date.
* Patients capable of providing informed consent before attending the first workshop

For carers

* Should be the primary carer nominated by a patient who fulfils the inclusion criteria, this includes parents of affected children
* Should be willing to participate in at least a 60-minute and ideally 90-minute workshops at the designated study location, time and date.
* Carers can only participate in the study with the cancer patient he/she is caring for. The patient has to also involved in the study
* Carers need to be capable of providing informed consent before attending the first workshop

For healthcare professionals

* All clinicians need to be current employees of the study site
* Doctors need to be employed at Specialist Registrar, Fellow or Consultant Level
* Nurses of all grades are invited to participate but ideally need to have had some involvement in the outpatient care of oncology patients

All participants:-

* Should be willing to have the session's recorded audio, transcripts and analysed data from the focus groups/workshops shared with Entia Ltd.
* should be willing to attend multiple 60 to 90 minute workshops.
* should be willing for photos and video footage to be taken during the interview.
* Participants attending workshops later in the development process must be comfortable consenting to finger prick testing/ assessing the ease of use of the test disposable

Exclusion Criteria:

For patients

* Does not have adequate English to participate in focus group interview without an interpreter
* Patients of the study site who are not currently undergoing systemic therapy or have previously undergone systemic therapy within the past 12 months
* Patients not willing to participate in at least 60-minute and ideally 90-minute focus group discussion at the designated study location, time and date.
* Participant not capable of providing consent or have a suitable, legally acceptable representative present to provide consent before the focus group interview.

For carers

* Is not the nominated primary carer of a cancer patient who fulfils the inclusion criteria, this includes parents of affected children
* Not paired with a patient that is involved in the study
* Carers not willing to participate in at least a 60-minute and ideally 90-minute focus group discussion at the designated study location, time and date.

For healthcare professionals

● Doctors who are not employed at Specialist Registrar, Fellow or Consultant Level

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Patients currently undergoing or who have previously undergone, systemic therapy within the past 12 months.
  * Carers of eligible patients.
  * Healthcare professionals and experts employed at the study sites. This will include:
    * Specialist registrars, fellows, consultants, nurses
    * Laboratory and Information Technology experts
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Qualitative capture of user feedback- focus groups | 30 months
  Participant feedback on the iterative designs of a future home-based monitoring service in order to arrive at a final prototype device and service design, suitable for patient, carer and healthcare professional's use.

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom